CLINICAL TRIAL: NCT04228042
Title: Tolerability and Activity of Neoadjuvant Infigratinib, an Inhibitor of FGFR, in Upper Tract Urothelial Carcinoma
Brief Title: Infigratinib Before Surgery for the Treatment of Upper Tract Urothelial Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Drug manufacturer made the business decision to cease all infigratinib oncology research in the US and withdrew the IND
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-0557; NCI-2019-08197 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2019-0557 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2019-12-30; First posted 2020-01-14 (Actual); Results first posted 2025-01-01 (Actual); Last update posted 2025-01-01 (Actual); Status verified 2024-09

CONDITIONS: Renal Pelvis and Ureter Urothelial Carcinoma
MeSH Terms: interventions — infigratinib; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (infigratinib, surgery) (Experimental): Patients receive infigratinib PO QD on days 1-21. Treatment repeats every 28 days for up to 2 cycles in the absence of disease progression or unacceptable toxicity. During weeks 8-9 (at least 48 hours after last dose of infigratinib), patients undergo surgery.
  Interventions: Drug: Infigratinib; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Procedure: Surgical Procedure

INTERVENTIONS:
Drug: Infigratinib — Given PO
  Other Names: 3-(2,6-Dichloro-3,5-dimethoxyphenyl)-1-(6-((4-(4-ethylpiperazin-1-yl)phenyl)amino)pyrimidin-4-yl)-1-methylurea; BGJ-398; BGJ398
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies
Procedure: Surgical Procedure — Undergo surgery
  Other Names: Operation; Surgery; Surgical; Surgical Intervention; Surgical Interventions; Surgical Procedures; Type of Surgery

SUMMARY:
This phase Ib trial studies the side effects of infigratinib before surgery in treating patients with upper tract urothelial cancer. Infigratinib may stop the growth of tumor cells by blocking the activities of a gene called FGFR needed for cell growth. Giving infigratinib before surgery may cause the tumor to shrink, which may make the surgical procedure easier and/or reduce the need for more extensive surgery.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Evaluate the tolerability of infigratinib in patients with low-grade and high-grade platinum ineligible upper tract urothelial carcinoma (UTUC).

SECONDARY OBJECTIVES:

I. Assess tolerability in those with GFR 30-49. II. Evaluate the objective response rate (complete response [CR] + partial response [PR]) of infigratinib after 2 cycles in UTUC with and without FGFR3 alterations.

III. Correlate tumor tissue FGFR3 alteration (presence/absence, alteration type, and clonal status) with response and occurrence/severity of adverse events (AEs) such as hyperphosphatemia.

IV. Evaluate upper tract, bladder and local/distant recurrence within 12 months.

V. Evaluate renal function pre-treatment and after two treatments. VI. Evaluate patient-reported quality of life (QOL) outcomes during treatment.

EXPLORATORY OBJECTIVES:

I. Explore intra-tumor heterogeneity, gene expression profiles, and changes in tumor microenvironment using single cell ribonucleic acid (RNA) sequencing (scRNA-seq) and mass cytometry by time-of-flight (CyTOF) pre and post treatment to identify potential mechanisms of response and/or resistance, and correlation with the occurrence/severity of AEs.

II. Explore urinary/upper tract washing FGFR3 alterations as potential biomarker for detection and response.

III. Explore cell free deoxyribonucleic acid (cfDNA) for detection of FGFR3 alterations and as a predictor of response.

OUTLINE:

Patients receive infigratinib orally (PO) once daily (QD) on days 1-21. Treatment repeats every 28 days for up to 2 cycles in the absence of disease progression or unacceptable toxicity. During weeks 8-9 (at least 48 hours after last dose of infigratinib), patients undergo surgery.

After completion of study treatment, patients are followed up at 30 days, then every 3 months for up to 1 year after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Have low grade UTUC undergoing nephroureterectomy or ureterectomy, or high grade UTUC and not eligible for cis-platin neoadjuvant chemotherapy either due to medical comorbidities (e.g., cardiac dysfunction, hearing loss, glomerular filtration rate [GFR] < 50), or based on < 49% risk prediction of non-organ confined disease by clinical nomogram
* Have adequate biopsy tissue available for mutational analysis, as determined by the study pathologist, prior to enrollment. Any biopsy of index UTUC tissue available within 6 weeks of enrollment may be used
* Calculated or measured creatinine clearance >= 30 mL/min
* Have an Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* Are able to read and/or understand the details of the study and provide written evidence of informed consent as approved by Institutional Review Board (IRB)/Independent Ethics Committee (IEC)
* Have recovered from AEs of previous systemic anti-cancer therapies to baseline or grade 1, except for alopecia
* Are able to swallow and retain oral medication
* Are willing and able to comply with scheduled visits, treatment plan and laboratory tests
* If a woman of childbearing potential (WOCBP), must have a negative pregnancy test within 7 days of the first dose of study drug. A woman is not of childbearing potential if she has undergone surgical sterilization (total hysterectomy, or bilateral tubal ligation or bilateral oophorectomy at least 6 weeks before taking study drug) or if she is post-menopausal and has had no menstrual bleeding of any kind including menstrual period, irregular bleeding, spotting, etc., for at least 12 months, with an appropriate clinical profile, and there is no other cause of amenorrhea (e.g., hormonal therapy, prior chemotherapy). WOCBP and males whose sexual partners are WOCBP must agree to use barrier contraception and a second form of highly effective contraception (Clinical Trials Facilitation Group, 2014) while receiving study drug and for 3 months following their last dose of study drug. Alternatively, total abstinence is also considered a highly effective contraception method when this is in line with the preferred and usual lifestyle of the subject. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception. Sexually active males must use a condom during intercourse while taking drug and for 3 months after the last dose of the study drug and should not father a child during this period. A condom is required to be used also by vasectomized men as well as during intercourse with a male partner to prevent delivery of the drug via seminal fluid

Exclusion Criteria:

* Have a history of another primary malignancy within 3 years except:

  * Adequately treated in situ carcinoma of the cervix, non-melanoma carcinoma of the skin
  * Any other untreated cancer deemed by treating physician to be at low risk for progression during the study period (such as low or intermediate risk prostate cancer)
  * Curatively treated malignancy that is not expected to have recurrence or require treatment during the course of the study
* Have uncontrolled bladder cancer. Patients with bladder cancer must have bladder cleared of disease by transurethral resection prior to initiating treatment and must not be at need for systemic therapy
* Have any other medical condition that would, in the investigator's judgment, prevent the subject's participation in the clinical study due to safety concerns or compliance with clinical study procedures
* Have current evidence of corneal or retinal disorder/keratopathy including, but not limited to, bullous/band keratopathy, corneal abrasion, inflammation/ulceration, keratoconjunctivitis, confirmed by ophthalmologic examination. Subjects with asymptomatic ophthalmologic conditions assessed by the investigator to pose minimal risk for study participation may be enrolled in the study
* Have a history and/or current evidence of extensive tissue calcification including, but not limited to, the soft tissue, kidneys, intestine, myocardium, vasculature and lung with the exception of calcified lymph nodes, minor pulmonary parenchymal calcifications, and asymptomatic coronary calcification
* Have impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of oral infigratinib (e.g., ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, small bowel resection)
* Have current evidence of endocrine alterations of calcium/phosphate homeostasis, e.g., parathyroid disorders, history of parathyroidectomy, tumor lysis, tumoral calcinosis etc
* Are currently receiving treatment with agents that are known strong inducers or inhibitors of CYP3A4 and medications which increase serum phosphorus and/or calcium concentration. Subjects are not permitted to receive enzyme-inducing anti-epileptic drugs, including carbamazepine, phenytoin, phenobarbital, and primidone
* Have consumed grapefruit, grapefruit juice, grapefruit hybrids, pomegranates, star fruits, pomelos, Seville oranges or products containing juice of these fruits within 7 days prior to first dose of study drug
* Have used medications known to prolong the QT interval and/or are associated with a risk of torsades de pointes (TdP) 7 days prior to first dose of study drug
* Have used amiodarone within 90 days prior to first dose of study drug
* Are currently using therapeutic doses of warfarin sodium or any other coumadin-derivative anticoagulants or using direct thrombin inhibitors (e.g., argatroban) or factor Xa inhibitors (e.g., rivaroxaban) that are primarily metabolized by CYP3A4. Heparin and/or low molecular weight heparins or direct thrombin inhibitors and/or factor Xa inhibitors that are not metabolized by CYP3A4 (e.g., dabigatran, edoxaban) are allowed
* Absolute neutrophil count (ANC) < 1,000/mm^3 (1.0 x 10^9/L)
* Platelets < 100,000/mm^3 (75 x 10^9/L)
* Hemoglobin < 9.0 g/dL
* Total bilirubin > 1.5 x upper limit of normal (ULN) (unless documented Gilbert's syndrome)
* Aspartate aminotransferase (AST)/ serum glutamic-oxaloacetic transaminase (SGOT) and alanine aminotransferase (ALT)/ serum glutamic-pyruvic transaminase (SGPT) > 2.5 x ULN (AST and ALT > 5 x ULN in the presence of liver involvement of cholangiocarcinoma)
* Calculated or measured creatinine clearance of < 30 mL/min
* Have amylase or lipase > 2.0 x ULN
* Have abnormal calcium-phosphate homeostasis:

  * Inorganic phosphorus outside of local normal limits
  * Total corrected serum calcium outside of local normal limits
* Have clinically significant cardiac disease including any of the following:

  * Congestive heart failure requiring treatment (New York Heart Association grade >= 2), left ventricular ejection fraction (LVEF) < 50% or local lower limit of normal as determined by echocardiogram (ECHO), or uncontrolled hypertension
  * Presence of Common Terminology Criteria for Adverse Events (CTCAE) version (v) 5.0 or later grade >= 2 ventricular arrhythmias, atrial fibrillation, bradycardia, or conduction abnormality
  * Unstable angina pectoris or acute myocardial infarction =< 3 months prior to first dose of study drug
  * Corrected QT interval by Fridericia (QTcF) > 470 msec (males and females)

    * Note: If the QTcF is > 470 msec in the first electrocardiography (ECG), a total of 3 ECGs separated by at least 5 minutes should be performed. If the average of these 3 consecutive results for QTcF is =< 470 msec, the subject meets eligibility in this regard
  * Known history of congenital long QT syndrome
* Have had a recent (=< 3 months) transient ischemic attack or stroke

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2020-07-28 (Actual); Primary Completion 2024-04-17 (Actual); Study Completion 2024-04-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mehrad Adibi, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was written to enroll and treat 20 participants, but enrollment was stopped because the drug manufacturer made the business decision to cease all infigratinib oncology research in the US and withdrew the IND that we cross-referenced in this IIT. Ultimately, 15 participants were consented, 1 patient screen failed, 14 completed the study
Groups:
- Infigratinib Plus Surgery: Patients will receive infigratinib 125 mg orally every day for a total of 2 cycles followed by surgery.
Period: Overall Study
Arm/Group | Infigratinib Plus Surgery
Started | 14
Completed | 14
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Infigratinib Plus Surgery
Number analyzed (Participants) | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 6
Age, Continuous [Median (Full Range); unit: years] | 63 [47 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 12
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 13
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability - TOX Rate
Description: The study will estimate percentage of patients who are not able to complete treatment (discontinuation) due to excessive toxicity along with the 90% exact confidence interval (NOTE: excessive toxicity is defined as treatment related adverse events that cause patients not to complete 2-cycles of planned treatment schedule, or delay in planned surgery greater than 14 days)
Time Frame: From day 1 until 30 days following last dose of infigratinib or until surgery, whichever occurs last, up to a total of 3 months.
Population: All patients who received at least one dose of infigratinib and completed surgery were included in the anlaysis. There were no delays to planned surgery in any of the participants
Measure: Number (90% Confidence Interval); unit: percentage of patients
Arm/Group | Infigratinib Plus Surgery
Number analyzed (Participants) | 14
percentage of patients | 14.30 [2.6 to 38.5]

2. Secondary Outcome: Evaluate the Objective Response Rate (CR+PR) of Infigratinib After 2 Cycles in UTUC With and Without FGFR3alterations
Description: Percentage of patients achieving a point in time objective response (either complete or partial response [CR or PR]) after 2 cycles of infigratinib. Tumor mapping will be performed from the endoscopic evaluation (after any biopsies) and this will be used to compare to pathologic (NUx/Ux cohort) or ureteroscopic (endoscopy cohort) findings in order to determine responses. Tumor mapping will be performed based on endoscopic findings, noting location, number of tumors, tumor architecture, and location of biopsies; and will again be performed during pathologic evaluation again noting size, location, number of tumors, architecture, and absence of tumor at any previously identified tumor. A difference of 3mm will be considered within error of measurement. All analyses will be performed on patients stratified as having or not having FGFR3 alterations.
Time Frame: Efficacy will be measured at time of surgery or approximately 2 months
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Infigratinib Plus Surgery
Number analyzed (Participants) | 14
percentage of participants | 66.7 [34.5 to 90.2]

3. Secondary Outcome: To Evaluate Patient-reported Quality of Life (QOL)
Description: Categorical variables were tabulated with frequency and percentage; continuous variables were summarized using descriptive statistics. A linear transformation to standardize the raw score was calculated for Functional/symptom scales and global health status (QOL) using the guidance in Scoring the EORTC QLQ-C30 version 3.0, so that scores range from 0 to 100. A higher score represents a higher ("better") level of functioning, or a higher ("worse") level of symptoms.
  Wilcoxon signed rank test was applied to compare functional/symptom scales and global health status (QOL) between different time points. A higher score for symptoms represents a worse outcome.
Time Frame: QoL surveys were obtained at baseline (day 1), pre-op after having received infigratinib for 2 cycles and 30 days after surgery, up to 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Infigratinib Plus Surgery
Number analyzed (Participants) | 14
score on a scale
  Fatigue score: Pre-OP | 17.46 (12.1)
  Fatigue score: post-OP | 15.08 (20.26)
  Score of diarrhea: At screening | 12.82 (21.68)
  Score of diarrhea: Pre-OP | 12.80 (16.88)
  Scores of appetite loss: At screening | 4.76 (12.1)
  Scores of appetite loss: Pre-OP | 19.05 (21.54)
  Scores of appetite loss: 30 days Post-OP | 7.14 (14.19)
Statistical Analysis 1: Comparison: Infigratinib Plus Surgery; Test type: Superiority; p = 0.009, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Infigratinib Plus Surgery; Test type: Superiority; p = 0.04, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Infigratinib Plus Surgery; Test type: Superiority; p = 0.003, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Infigratinib Plus Surgery; Test type: Superiority; p = 0.03, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: From day 1 until 30 days following last dose of infigratinib or until surgery, whichever occurs last, up to a total of 3 months.
Arm/Group | Infigratinib Plus Surgery
All-Cause Mortality (participants affected / at risk) | 0/14
Serious Adverse Events (participants affected / at risk) | 1/14
Other Adverse Events (participants affected / at risk) | 12/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Infigratinib Plus Surgery (N=14)
Hyponatremia (Investigations) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Infigratinib Plus Surgery (N=14)
Hyperphosphatemia (Investigations) | 9 (9)
Hyponatremia (Investigations) | 2 (2)
Lipase Increase (Investigations) | 3 (3)
Amylase Increase (Investigations) | 2 (2)
Hyperkalemia (Investigations) | 2 (2)
Creatinine Increase (Investigations) | 2 (2)
BUN Increase (Investigations) | 1 (1)
Cytokine Release Syndrome (Investigations) | 1 (1)
Anemia (Investigations) | 1 (1)
Hypercalcemia (Investigations) | 1 (1)
Hypophosphatemia (Investigations) | 1 (1)
WBC Decreased (Investigations) | 1 (1)
ALT Increase (Investigations) | 2 (2)
AST Increase (Investigations) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 7 (7)
Constipation (Gastrointestinal disorders) | 5 (5)
Disgeusia (Gastrointestinal disorders) | 5 (5)
Anorexia (Metabolism and nutrition disorders) | 3 (3)
Dry Mouth (Skin and subcutaneous tissue disorders) | 3 (3)
Nausea (Gastrointestinal disorders) | 1 (1)
Stomatitis/Sore throat (Skin and subcutaneous tissue disorders) | 1 (1)
Xerostomy (Skin and subcutaneous tissue disorders) | 1 (1)
Dry Eyes (Skin and subcutaneous tissue disorders) | 3 (3)
Blurred Vision (Skin and subcutaneous tissue disorders) | 1 (1)
Eye Pain (Skin and subcutaneous tissue disorders) | 1 (1)
Pingueculitis (Skin and subcutaneous tissue disorders) | 1 (1)
Sub-retinal Fluid (Skin and subcutaneous tissue disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 3 (3)
Nail Infection (Skin and subcutaneous tissue disorders) | 3 (3)
Skin Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Palmar-Plantar Erythrodysesthesia (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Fatigue (Investigations) | 4 (4)
Jaw Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Flank Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Headache (General disorders) | 1 (1)
Epistaxis (Skin and subcutaneous tissue disorders) | 3 (3)
Hematuria (Renal and urinary disorders) | 1 (1)
Lightheadedness (General disorders) | 1 (1)
Lower Leg Edema (Blood and lymphatic system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-09-23): https://cdn.clinicaltrials.gov/large-docs/42/NCT04228042/Prot_SAP_000.pdf